CLINICAL TRIAL: NCT01870401
Title: A Prospective, Multicenter, Single Blind, Randomized, Controlled Trial Comparing the Lutonix Drug Coated Balloon Versus Standard Balloon Angioplasty for Treatment of Below-the-Knee (BTK) Arteries(Lutonix BTK Trial)
Brief Title: Lutonix DCB Versus Standard Balloon Angioplasty for Treatment of Below-The-Knee (BTK) Arteries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Collaborators: Bard Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CL0005-01
Record Dates: First submitted 2013-05-07; First posted 2013-06-06 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Lutonix DCB (Experimental): Lutonix Paclitaxel Drug Coated Balloon
  Interventions: Device: Lutonix DCB
- PTA Catheter (Active Comparator): Standard Uncoated PTA Catheter
  Interventions: Device: Uncoated PTA Catheter

INTERVENTIONS:
Device: Lutonix DCB
  Other Names: LTX DCB
  Arms: Lutonix DCB
Device: Uncoated PTA Catheter
  Other Names: PTA
  Arms: PTA Catheter

SUMMARY:
To assess the safety and efficacy of the Lutonix Drug Coated Balloon (DCB) for treatment of stenosis or occlusion of native below-the-knee arteries.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female ≥18 years of age;
* Rutherford Clinical Category 3, 4 & 5;
* Life expectancy ≥ 1 year;
* Significant stenosis (≥70%)
* A patent inflow artery;
* Target vessel(s) diameter between 2 and 4 mm;
* Target vessel(s) reconstitute(s) at or above the ankle

Exclusion Criteria:

* Pregnant or planning on becoming pregnant;
* History of stroke within 3 months;
* History of MI, thrombolysis or angina within 30 days of enrollment;
* Planned major amputation (of either leg)
* Prior major amputation if amputation occurred less than one year prior to enrollment and if patient is not independently ambulating;
* GFR ≤ 30 ml/min per 1.73m2;
* Acute limb ischemia;
* In-stent restenosis of target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Geraghty, MD, Principal Investigator — Washington University School of Medicine; Jihad Mustapha, MD, Principal Investigator — Metro Health Hospital; Marianne Brodmann, MD, Principal Investigator — Medical University Graz, Austria
Locations (51):
- United States (33):
  - Yale University-Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Cardiovascular Solutions Institute, LLC, Bradenton, Florida
  - Morton Plant Mease Health Care, Inc, Clearwater, Florida
  - Cardiovascular Research of North Florida, LLC, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Radiology and Imaging Specialists of Lakeland, P.A, Lakeland, Florida
  - Mt. Sinai Medical Center, Miami Beach, Florida
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Central Iowa Hospital Corporation, West Des Moines, Iowa
  - CIS Clinical Research Corporation, Houma, Louisiana
  - Steward St. Elizabeth Medical Center of Boston, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Metro Health-University of Michigan Health Hospital, Wyoming, Michigan
  - Jackson Heart Clinic, P.A., Jackson, Mississippi
  - Barnes Jewish Hospital, St Louis, Missouri
  - Deborah Heart & Lung Ctr, Browns Mills, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New Mexico Heart Institute, LLC, Albuquerque, New Mexico
  - Mount Sinai School of Medicine, New York, New York
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - Trihealth Heart Institute, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Corporation, Columbus, Ohio
  - Providence Health & Service - Oregon, Portland, Oregon
  - The Miriam Hospital - A Lifespan Partner, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University Surgical Associates, LLC, Chattanooga, Tennessee
  - Wellmont Cardiology Services, Inc., Kingsport, Tennessee
  - Austin Heart PLLC, Austin, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - Charleston Area Medical Center Health System, Charleston, West Virginia
  - Aurora St. Luke's Vascular Center, Milwaukee, Wisconsin
- Medical University Graz, Graz, Austria
- ZOL St. Jan, Genk, Belgium
- University Health Network, Toronto, Ontario, Canada
- Germany (8):
  - Klinik für Kardiologie • Klinikum Arnsberg GmbH, Arnsberg
  - Universitaets Herzzentrum Freiburg/Bad Krozingen, Bad Krozingen
  - Med. Universitaet Heidelberg,Herzzentrum (Abteilung Innere Medizin III), Heidelberg
  - Hospital Kempten, Immenstadt im Allgäu
  - Universitaetsklinikum Leipzig Medical Centre, Leipzig
  - Universitätsklinikum Münster, Innere Medizin C, Münster
  - Medinos Kliniken des Landkriess Sonneberg GmbH, Sonneberg
  - University of Tubingen, Dept. of Diagnostic and Interventional Radiology, Tübingen
- Maria Cecilia Hospital, Cotignola, Italy
- Japan (5):
  - Kasukabe Chuo General Hospital, Kasukabe
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Morinomiya Hospital, Osaka
  - Kishiwada Tokushukai Hospital, Osaka
  - Toho University, Tokyo
- Kantonsspital Luzern, Lucerne, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from medical clinics and hospitals between June 2013 and January 2018. The first participant was enrolled on June 3, 2013 and the last participant enrolled was on December 12, 2017.
Groups:
- Lutonix DCB: Percutaneous transluminal angiography (PTA) will be performed using the Lutonix Drug Coated Balloon.
  Lutonix DCB
  Percutaneous Transluminal Angiography: Percutaneous transluminal angioplasty (PTA) is a procedure that can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored.
- Standard Balloon Angioplasty Catheter: Percutaneous transluminal angiography (PTA) will be performed using a commercially available uncoated PTA balloon. Balloons with an external wire support, cutting/scoring component or other similar modifications are not permitted. Multiple balloons, inflations and/or prolonged inflation may be used.
  Standard Balloon Angioplasty Catheter
  Percutaneous Transluminal Angiography: Percutaneous transluminal angioplasty (PTA) is a procedure that can open up a blocked blood vessel using a small, flexible plastic tube, or catheter, with a "balloon" at the end of it. When the tube is in place, it inflates to open the blood vessel, or artery, so that normal blood flow is restored.
Period: Overall Study
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Started | 287 | 155
Completed | 137 | 59
Not Completed | 150 | 96
Not completed — Death | 48 | 24
Not completed — Withdrawal by Subject | 39 | 26
Not completed — Lost to Follow-up | 19 | 14
Not completed — Other | 9 | 7
Not completed — On-going in the Study | 35 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter | Total
Number analyzed (Participants) | 287 | 155 | 442
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (9.65) | 72.9 (9.62) | 72.9 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 51 | 136
  Male | 202 | 104 | 306
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 25 | 15 | 40
  Black or African American | 33 | 12 | 45
  White | 226 | 127 | 353
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 178 | 97 | 275
  Europe | 80 | 42 | 122
  Japan | 25 | 15 | 40
  Canada | 4 | 1 | 5
Weight [Mean (Standard Deviation); unit: kg] | 82.6 (21.15) | 81.9 (20.29) | 82.3 (20.83)
Height [Mean (Standard Deviation); unit: cm] | 170 (10.07) | 170 (10.65) | 170 (10.26)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (6.31) | 28.0 (5.65) | 28.2 (6.08)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Below-the-Knee (BTK) Major Adverse Limb Event and Peri-Operative Death (POD) at 30 Days Post Index Procedure.
Description: The primary safety endpoint is defined as freedom from the composite of all-cause death, above-ankle amputation or major reintervention (new bypass graft, jump/interposition graft revision, or thrombectomy/thrombolysis) of the index limb involving a below-the-knee artery.
Time Frame: 30 days post index procedure
Population: The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Lutonix DCB: Lutonix Paclitaxel Drug Coated Balloon
  Lutonix DCB
- PTA Catheter: Standard Uncoated PTA Catheter
  Uncoated PTA Catheter
Arm/Group | Lutonix DCB | PTA Catheter
Number analyzed (Participants) | 286 | 155
Participants | 284 | 154
Statistical Analysis 1: Comparison: Lutonix DCB vs PTA Catheter; The primary safety hypothesis is as follows: H0: pControl - pDCB ≥ and H1: pControl (alpha) pDCB < where p is the success rate in each arm and (alpha) is the non-inferiority bound; Test type: Non-Inferiority — The protocol identified a non-inferiority bound equal to 0.12 (12%); p < 0.025, Farrington and Manning

2. Primary Outcome: Number of Participants With Freedom From the Composite of Above-ankle Amputation, Target Lesion Occlusion, and Clinically-driven Target Lesion Revascularization at 6 Months Post Index Procedure.
Description: The primary efficacy endpoint is defined as freedom from the composite of above-ankle amputation, target lesion occlusion, and clinically-driven target lesion revascularization. All amputations included in endpoints refer to amputations in the index limb.
Time Frame: 6 months post-index procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 269 | 137
Participants | 201 | 88
Statistical Analysis 1: Comparison: Lutonix DCB vs Standard Balloon Angioplasty Catheter; Test type: Superiority; p = 0.0222, Wald Test; One-sided Wald test based on model estimate of DCB treatment effect and subject as a random effect

3. Secondary Outcome: Percentage of Lesions Considered Technical Success at Time of Index Procedure
Description: Technical Success: A success is determined if the device success was achieved and a final residual stenosis post study device (DCB or placebo) dilatation ≤ 30% was reported.
Time Frame: At time of index procedure
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Lesions) | 106 | 60
percentage of lesions | 61.3 [51.4 to 70.6] | 58.3 [44.9 to 70.9]

4. Secondary Outcome: Percentage of Procedures With Procedural Success at Time of Index Procedure.
Description: A success is determined if there is restoration of at least 1 infrapopliteal artery with residual stenosis ≤ 30% (or ≤ 50% depending upon the version of the protocol) and inline outflow to the foot, irrespective of device success, and without a major adverse event during the index procedure.
Time Frame: At time of Index Procedure
Measure: Number (95% Confidence Interval); unit: Percentage of Procedures
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Percentage of Procedures | 84.0 [79.5 to 87.9] | 81.4 [74.8 to 86.8]

5. Secondary Outcome: Comparison of the Below the Knee (BTK) Major Adverse Limb Event (MALE) and Perioperative Death (POD) Rate to a Performance Goal at 30 Days Post Index Procedure.
Time Frame: 30 days post index procedure
Population: Data were not collected.
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in European Quality of Life 5 Dimensions (EuroQol -5D) Scores at 30 Days, 6 and 12 Months Compared to Baseline.
Description: Mean change in EuroQol (EQ-5D) scores at 30 days, 6, and 12 months compared to baseline. The EurolQol-5D system rates quality of life using five dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels of ratings, that is, no problems, slight problems, moderate problems, severe problems and extreme problems that can be selected. A visual scale allows participants to report their own perception of their health status. The overall scores range from 0 (worst) to 100 (best). Please note that the data in the table below represent the mean changes in overall scores for each group compared to their baseline data. Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure compared to baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Scores on a scale
  30-days Post Index Procedure: number analyzed (Participants) | 33 | 20
  30-days Post Index Procedure | 1.10 (0.458) | 0.53 (0.533)
  6 months post index procedure: number analyzed (Participants) | 245 | 125
  6 months post index procedure | 0.07 (0.300) | 0.05 (0.297)
  12 months post index procedure: number analyzed (Participants) | 227 | 114
  12 months post index procedure | 0.09 (0.284) | 0.12 (0.267)

7. Secondary Outcome: Late Lumen Loss at 12 Months Post Index Procedure
Time Frame: 12 months post-index procedure
Population: Data were not collected.
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Healed Wounds at 30 Days, 6 and 12 Months Post Index Procedure
Description: Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available. The number of wounds analyzed at 6 and 12 months post-index procedure includes wounds that may have appeared (new wounds) since the previous time period reporting.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: as for outcome 1
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Wounds) | 211 | 114
Wounds
  30-days Post Index Procedure: number analyzed (Participants) | 287 | 143
  30-days Post Index Procedure | 49 | 24
  6 months post index procedure: number analyzed (Participants) | 287 | 122
  6 months post index procedure: number analyzed (Wounds) | 166 | 82
  6 months post index procedure | 61 | 45
  12 months post index procedure: number analyzed (Participants) | 287 | 108
  12 months post index procedure: number analyzed (Wounds) | 103 | 55
  12 months post index procedure | 42 | 17

9. Secondary Outcome: Number of Non-Healed Wounds by Category (Improving, Stagnant and Worsening) at 30 Days, 6 and 12 Months Post-Index Procedure.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: as for outcome 1
Measure: Count of Units; unit: Non-Healed Wounds
Units Other Than Participants: Non-Healed Wounds
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Non-Healed Wounds) | 130 | 61
Non-Healed Wounds
  30-days Post Index Procedure: Improving | 90 | 37
  30-days Post Index Procedure: Stagnant | 24 | 16
  30-days Post Index Procedure: Worsening | 16 | 8
  6 months post index procedure: number analyzed (Non-Healed Wounds) | 51 | 17
  6 months post index procedure: Improving | 26 | 6
  6 months post index procedure: Stagnant | 13 | 7
  6 months post index procedure: Worsening | 12 | 4
  12 months post index procedure: number analyzed (Non-Healed Wounds) | 28 | 14
  12 months post index procedure: Improving | 18 | 8
  12 months post index procedure: Stagnant | 9 | 4
  12 months post index procedure: Worsening | 1 | 2

10. Secondary Outcome: Percentage of Existing, New, and Recurrent Wounds at 30 Days, 6 and 12 Months Post Index Procedure.
Description: Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: Participants may have more than one wound type or wounds in more than one location. The number of participants (n) varies from the total number of participants (N) in the study as n depends on the number of participants for which data was available at the given time-point analysis.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 178 | 97
Number analyzed (Wounds) | 100 | 67
Wounds
  30-days Post Index Procedure: number analyzed (Wounds) | 100 | 58
  30-days Post Index Procedure: Existing Wounds | 94 | 46
  30-days Post Index Procedure: New Wounds | 5 | 12
  30-days Post Index Procedure: Recurrent Wounds | 1 | 0
  6 months post index procedure: number analyzed (Wounds) | 83 | 44
  6 months post index procedure: Existing Wounds | 62 | 33
  6 months post index procedure: New Wounds | 20 | 10
  6 months post index procedure: Recurrent Wounds | 1 | 1
  12 months post index procedure: number analyzed (Wounds) | 50 | 26
  12 months post index procedure: Existing Wounds | 37 | 16
  12 months post index procedure: New Wounds | 9 | 9
  12 months post index procedure: Recurrent Wounds | 4 | 1

11. Secondary Outcome: Change in Rutherford Classification Scores at 30 Days, 6 and 12 Months Post Index Procedure Compared to Baseline.
Description: The endpoint summarizes the change in index-limb Rutherford Classification of participants from baseline through 36 months. Data is presented as shift from baseline Rutherford Classification data using the following categories: 1) Improvement, 2) Same, and 3) Worsened.
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure compared to baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Participants
  30-days Post Index Procedure: number analyzed (Participants) | 263 | 144
  30-days Post Index Procedure: Improved | 161 | 83
  30-days Post Index Procedure: Same | 100 | 59
  30-days Post Index Procedure: Worsened | 2 | 2
  6 months post index procedure: number analyzed (Participants) | 243 | 120
  6 months post index procedure: Improved | 179 | 98
  6 months post index procedure: Same | 58 | 21
  6 months post index procedure: Worsened | 6 | 1
  12 months post index procedure: number analyzed (Participants) | 220 | 110
  12 months post index procedure: Improved | 176 | 90
  12 months post index procedure: Same | 39 | 16
  12 months post index procedure: Worsened | 5 | 4

12. Secondary Outcome: Number of Participants With Freedom From Above Ankle Amputation, Unhealed Wound, Ischemic Rest Pain, Target Vessel Occlusion, and Clinically-Driven Target Vessel Revascularization (TVR) at 30 Days, 6 and 12 Months Post Index Procedure.
Description: The composite endpoint of freedom from above ankle amputation (CEC-adjudicated), unhealed wound (presence of wound vs. no wound), ischemic rest pain (Rutherford category 4 or higher), target vessel occlusion (based on DUS and/or angiograph), and clinically-driven TVR (CEC-adjudicated).
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Participants
  30-days Post Index Procedure: number analyzed (Participants) | 263 | 140
  30-days Post Index Procedure | 98 | 49
  6 months post index procedure: number analyzed (Participants) | 241 | 126
  6 months post index procedure | 93 | 45
  12 months post index procedure: number analyzed (Participants) | 224 | 118
  12 months post index procedure | 71 | 53

13. Secondary Outcome: Percentage of Participants With Freedom From Primary Patency Failure at 30 Days, 6 and 12 Months Post Index Procedure
Description: Primary patency is defined as the absence of both total occlusion (100% diameter stenosis) in all of the target lesions in a flow pathway as well as a clinically-driven Target Lesion Revascularization (TLR).
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days and at 6 and 12 months
Population: The number of participants or lesions may vary depending on the number of participants/lesions for which data was available at the given time-point analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 261 | 127
Percentage of Participants
  30-days Post Index Procedure | 97.4 [94.6 to 98.7] | 94.8 [89.4 to 97.5]
  6 months post index procedure: number analyzed (Participants) | 208 | 85
  6 months post index procedure | 85.3 [80.2 to 89.1] | 72.2 [63.3 to 79.3]
  12 months post procedure: number analyzed (Participants) | 127 | 66
  12 months post procedure | 58.1 [51.5 to 64.2] | 60.0 [50.6 to 68.2]

14. Secondary Outcome: Percentage of Lesions With Primary Patency Excluding Early Mechanical Recoil at 30 Days, 6 and 12 Months Post Index Procedure
Description: Primary patency with exclusion of early mechanical recoil of the target flow pathway is defined as the absence of both total occlusion (100% diameter stenosis) of the target lesions and clinically-driven TLR events > 30 days.
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of Lesions
Units Other Than Participants: Lesions
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Lesions) | 298 | 159
Percentage of Lesions
  30-days Post Index Procedure | 100 [100 to 100] | 100 [100 to 100]
  6 months post index procedure: number analyzed (Lesions) | 237 | 99
  6 months post index procedure | 88.0 [83.5 to 91.3] | 73.8 [65.5 to 80.4]
  12 months post index procedure: number analyzed (Lesions) | 151 | 78
  12 months post index procedure | 61.7 [55.4 to 67.3] | 63.0 [54.2 to 70.6]

15. Secondary Outcome: Number of Lesions With Secondary Patency at 30 Days, 6 and 12 Months Post Index Procedure
Description: The secondary patency of the target lesion is defined as the absence of total occlusion (100% diameter stenosis) of the target lesions based on angiography (if performed) or ultrasound as analyzed by the angiographic Core Lab.
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: as for outcome 1
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Lesions) | 293 | 184
Lesions
  30-days Post Index Procedure: number analyzed (Lesions) | 293 | 155
  30-days Post Index Procedure | 284 | 146
  6 months post index procedure: number analyzed (Lesions) | 259 | 126
  6 months post index procedure | 217 | 103
  12 months post index procedure: number analyzed (Lesions) | 213 | 110
  12 months post index procedure | 144 | 91

16. Secondary Outcome: Composite of Freedom From Clinically -Driven Target Lesion Revascularization (TLR) and From 50% DS by Angiography or Duplex Ultrasound at 30 Days, 6 and 12 Months Post Index Procedure.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: Data were not collected.
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change in Toe Brachial Index (TBI) at 30 Days, 6 and 12 Months Post Index Procedure Compared to Baseline
Description: Mean change from baseline values. The Toe Brachial Index (TBI) is defined as a ratio of toe to brachial (upper arm) artery systolic blood pressure and aims at determining how well the blood is flowing in the legs.
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure compared to baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 119 | 128
Ratio
  30-days Post Index Procedure | 0.20 (0.25) | 0.28 (0.42)
  6 months post index procedure: number analyzed (Participants) | 104 | 113
  6 months post index procedure | 0.15 (0.24) | 0.17 (0.43)
  12 months post index procedure: number analyzed (Participants) | 84 | 104
  12 months post index procedure | 0.12 (0.23) | 0.18 (0.40)

18. Secondary Outcome: Change in Ankle Brachial Index (ABI) at 30 Days, 6 and 12 Months Post Index Procedure Compared to Baseline
Description: Mean change from baseline values. The Ankle Brachial Index (ABI) is defined as a ratio of ankle to brachial (upper arm) artery systolic blood pressure and aims at determining how well the blood is flowing in the legs.
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, and at 6 and 12 months compared to baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 237 | 128
Ratio
  30-days Post Index Procedure | 0.23 (0.36) | 0.28 (0.42)
  6 months post index procedure: number analyzed (Participants) | 218 | 113
  6 months post index procedure | 0.16 (0.36) | 0.17 (0.43)
  12 months post index procedure: number analyzed (Participants) | 193 | 104
  12 months post index procedure | 0.11 (0.36) | 0.18 (0.40)

19. Secondary Outcome: Change in Walking Impairment Questionnaire (WIQ) Scores at 30 Days, 6 and 12 Months Post Index Procedure Compared to Baseline.
Description: The WIQ assesses 3 categories of activities that include 1) walking distance, 2) stair-climbing, and 3) walking speed. Each question requires participants to rate their degree of difficulty with the activity on a scale of 0 (unable) to 4 (no problem). Final scores range from 0% to 100%, with lower percentages indicating higher levels of difficulties with activities.The results below represent the mean differences in total Walking Impairment Questionnaire (WIQ) scores at 30 days 6 and 12 months, compared to baseline assessment scores.
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure compared to baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 238 | 120
score on a scale
  30-days Post Index Procedure: number analyzed (Participants) | 221 | 117
  30-days Post Index Procedure | 0.3 (18.13) | 1.1 (17.46)
  6 months post index procedure | 2.9 (21.55) | 3.6 (20.27)
  12 months post index procedure: number analyzed (Participants) | 218 | 110
  12 months post index procedure | 2.7 (22.10) | 2.3 (20.23)

20. Secondary Outcome: Number of Participants With Clinically-Driven Target Lesion Revascularization (TLR) at 30 Days, 6 and 12 Months Post Index Procedure
Time Frame: 30 days, 6 and 12 months post index procedure
Population: Data were not collected.
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Cumulative Number of Target Lesion Revascularization (TLR) at 30 Days, 6 and 12 Months Post Index Procedure.
Description: Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Measure: Number; unit: participants
Units Other Than Participants: Target Lesions Revascularization
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Target Lesions Revascularization) | 170 | 75
participants
  30-days Post Index Procedure | 5 | 6
  6 months post index procedure | 36 | 36
  12 months post index procedure | 101 | 53

22. Secondary Outcome: Number of Participants With Clinically-Driven Target Vessel Revascularization (TVR) at 30 Days, 6 and 12 Months Post Index Procedure.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: Data were not collected.
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Cumulative Number of Target Vessel Revascularization (TVR) at 30 Days, 6 and 12 Months Post Index Procedure.
Time Frame: 30 days, 6 and 12 months post index procedure
Measure: Number; unit: Target Vessel Revascualarization
Units Other Than Participants: Target Vessel Revascularization
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Target Vessel Revascularization) | 175 | 79
Target Vessel Revascualarization
  30-days Post Index Procedure | 5 | 6
  6 months post index procedure | 37 | 38
  12 months post index procedure | 105 | 57

24. Secondary Outcome: Percentage of Participants With Freedom From Limb Amputation at 30 Days, 6 and 12 Months Post Index Procedure
Description: Limb salvage defined as no amputation of target limb.
Time Frame: 30 days and at 6 and 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 282 | 153
percentage of participants
  30-days Post Index Procedure | 100 [100 to 100] | 100 [100 to 100]
  6 months post index procedure: number analyzed (Participants) | 266 | 138
  6 months post index procedure | 98.9 [96.6 to 99.6] | 98.0 [93.9 to 99.4]
  12 months post index procedure: number analyzed (Participants) | 241 | 125
  12 months post index procedure | 97.4 [94.5 to 98.7] | 98.0 [93.9 to 99.4]

25. Secondary Outcome: Percentage of Participants With Freedom From Unplanned Below the Knee (BTK) Amputation of the Target Limb at 30 Days, 6 and 12 Months Post Index Procedure.
Description: Defined as amputation that was below the ankle, including digit amputation. Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 274 | 148
Percentage of participants
  30-days Post Index Procedure | 95.8 [92.7 to 97.6] | 95.5 [90.8 to 97.8]
  6 months post index procedure: number analyzed (Participants) | 242 | 129
  6 months post index procedure | 88.6 [84.2 to 91.8] | 88.2 [81.9 to 92.4]
  12 months post index procedure: number analyzed (Participants) | 219 | 110
  12 months post index procedure | 86.3 [81.6 to 89.8] | 83.1 [76.0 to 88.3]

26. Secondary Outcome: Cumulative Number of of Below the Knee (BTK) Index-Limb Reinterventions at 30 Days, 6 and 12 Months Post Index Procedure.
Description: The overall burden of BTK reinterventions was defined as the total number of BTK index-limb re-interventions and major amputations for each time point.
  Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Measure: Number; unit: Limb Reintervention
Units Other Than Participants: Limb Reintervention
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Number analyzed (Limb Reintervention) | 365 | 164
Limb Reintervention
  30-days Post Index Procedure | 27 | 22
  6 months post index procedure | 112 | 88
  12 months post index procedure | 235 | 124

27. Secondary Outcome: Percentage of Participants With Freedom From Composite of Perioperative Death (POD), Index Limb-related Death, Below the Knee Reinterventions or Major Amputations of the Index Limb at 30 Days, 6 and 12 Months Post Index Procedure
Description: Results for 24 and 36 months will be reported when the final Clinical Study Report becomes available.
Time Frame: 30 days, 6 and 12 months post index procedure
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
Number analyzed (Participants) | 287 | 155
Percentage of participants
  30-days Post Index Procedure: number analyzed (Participants) | 267 | 140
  30-days Post Index Procedure | 93.4 [89.8 to 95.7] | 90.3 [84.5 to 94.0]
  6 months post index procedure: number analyzed (Participants) | 216 | 102
  6 months post index procedure | 78.9 [73.6 to 83.2] | 69.6 [61.6 to 76.3]
  12 months post index procedure: number analyzed (Participants) | 143 | 75
  12 months post index procedure | 56.8 [50.6 to 62.5] | 58.0 [49.5 to 65.6]

ADVERSE EVENTS:
Time Frame: Subjects with Serious Adverse Events by Body System and Preferred Term are presented through 36 Months and are Site-reported. All devices and procedure-related adverse events (AEs) were collected through 36 months post index procedure and are CEC adjudicated.
Arm/Group | Lutonix DCB | Standard Balloon Angioplasty Catheter
All-Cause Mortality (participants affected / at risk) | 48/287 | 25/155
Serious Adverse Events (participants affected / at risk) | 240/287 | 126/155
Other Adverse Events (participants affected / at risk) | 106/287 | 45/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lutonix DCB (N=287) | Standard Balloon Angioplasty Catheter (N=155)
Anaemia (Blood and lymphatic system disorders) | 10 | 3
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 1 | 0
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 3 | 1
Acute Myocardial Infarction (Cardiac disorders) | 14 | 8
Angina Pectoris (Cardiac disorders) | 8 | 6
Angina Unstable (Cardiac disorders) | 5 | 0
Aortic Valve Disease (Cardiac disorders) | 1 | 0
Aortic Valve Stenosis (Cardiac disorders) | 5 | 2
Arrhythmia Supraventricular (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 10 | 6
Atrial Flutter (Cardiac disorders) | 0 | 2
Atrial Tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular Block (Cardiac disorders) | 1 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Atrioventricular Block Second Degree (Cardiac disorders) | 2 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bundle Branch Block Left (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 4 | 2
Cardiac Failure (Cardiac disorders) | 11 | 5
Cardiac Failure Acute (Cardiac disorders) | 5 | 1
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 21 | 12
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 1
Coronary Artery Disease (Cardiac disorders) | 11 | 5
Coronary Artery Stenosis (Cardiac disorders) | 3 | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 6 | 2
Left Ventricular Failure (Cardiac disorders) | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 1 | 2
Myocardial Infarction (Cardiac disorders) | 2 | 2
Myocardial Ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Pulseless Electrical Activity (Cardiac disorders) | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 0 | 1
Sick Sinus Syndrome (Cardiac disorders) | 3 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Tricuspid Valve Disease (Cardiac disorders) | 1 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 2 | 0
Buried Penis Syndrome (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Angle Closure Glaucoma (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 1
Diabetic Retinopathy (Eye disorders) | 1 | 0
Eye Haemorrhage (Eye disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecal Incontinence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 7 | 2
Gastrointestinal Oedema (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 2 | 0
Intestinal Mass (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Ischaemic Enteritis (Gastrointestinal disorders) | 0 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 1
Mesenteric Artery Stenosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Adverse Drug Reaction (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 1
Death (General disorders) | 8 | 1
Device Battery Issue (General disorders) | 1 | 0
Device Dislocation (General disorders) | 0 | 2
Device Occlusion (General disorders) | 1 | 1
Disease Progression (General disorders) | 4 | 0
Impaired Healing (General disorders) | 8 | 3
Local Swelling (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0
Oedema Peripheral (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 4 | 0
Vessel Puncture Site Haematoma (General disorders) | 1 | 0
Vessel Puncture Site Haemorrhage (General disorders) | 2 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Abscess Limb (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 1
Arthritis Bacterial (Infections and infestations) | 2 | 0
Atypical Pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 5 | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 13 | 6
Clostridium Difficile Colitis (Infections and infestations) | 1 | 2
Clostridium Difficile Infection (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 0 | 2
Diabetic Foot Infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Emphysematous Cystitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 22 | 11
Gastritis Viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Groin Abscess (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 1
Infected Skin Ulcer (Infections and infestations) | 3 | 0
Influenza (Infections and infestations) | 2 | 0
Intervertebral Discitis (Infections and infestations) | 1 | 2
Localised Infection (Infections and infestations) | 10 | 5
Lung Abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 21 | 16
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 15 | 7
Pneumonia Bacterial (Infections and infestations) | 0 | 2
Postoperative Wound Infection (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 8 | 5
Septic shock (Infections and infestations) | 2 | 3
Serratia Bacteraemia (Infections and infestations) | 1 | 0
Sputum Purulent (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 9 | 6
Urosepsis (Infections and infestations) | 1 | 2
Vaginal Infection (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 8 | 2
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 | 1
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 3 | 0
Iatrogenic Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 35 | 11
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 62 | 36
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 2
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 3 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 2 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular Graft Complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 | 0
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 | 2
Wound (Injury, poisoning and procedural complications) | 15 | 6
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wound Necrosis (Injury, poisoning and procedural complications) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Blood Culture Positive (Investigations) | 1 | 0
Blood Glucose Fluctuation (Investigations) | 1 | 0
Blood Pressure Decreased (Investigations) | 1 | 0
Haemoglobin Decreased (Investigations) | 1 | 1
Investigation (Investigations) | 0 | 1
Radioisotope Scan Abnormal (Investigations) | 1 | 0
Troponin Increased (Investigations) | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 3 | 2
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0
Joint Contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft Tissue Mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenosquamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Brain Stem Stroke (Nervous system disorders) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 4 | 3
Carpal Tunnel Syndrome (Nervous system disorders) | 3 | 0
Cerebral Haemorrhage (Nervous system disorders) | 2 | 1
Cerebral Infarction (Nervous system disorders) | 5 | 1
Cerebrovascular Accident (Nervous system disorders) | 6 | 3
Cerebrovascular Disorder (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Embolic Stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 3 | 2
Hemiparesis (Nervous system disorders) | 1 | 0
Lacunar Infarction (Nervous system disorders) | 1 | 0
Metabolic Encephalopathy (Nervous system disorders) | 1 | 0
Parkinson's Disease (Nervous system disorders) | 2 | 0
Precerebral Artery Occlusion (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 6 | 1
Toxic Encephalopathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 0
Vascular Dementia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 5 | 2
Neglect Of Personal Appearance (Psychiatric disorders) | 1 | 0
Bladder Mass (Renal and urinary disorders) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 2
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy Toxic (Renal and urinary disorders) | 1 | 0
Obstructive Uropathy (Renal and urinary disorders) | 0 | 1
Pyuria (Renal and urinary disorders) | 0 | 1
Renal Artery Stenosis (Renal and urinary disorders) | 2 | 0
Renal Failure (Renal and urinary disorders) | 10 | 7
Renal Failure Acute (Renal and urinary disorders) | 12 | 3
Renal Impairment (Renal and urinary disorders) | 1 | 0
Ureteric Stenosis (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 | 1
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Dry Gangrene (Skin and subcutaneous tissue disorders) | 0 | 2
Leukocytoclastic Vasculitis (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 3 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 17 | 12
Accelerated Hypertension (Vascular disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1
Aortic Stenosis (Vascular disorders) | 2 | 0
Arterial Rupture (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 6 | 2
Diabetic Macroangiopathy (Vascular disorders) | 1 | 0
Embolism Arterial (Vascular disorders) | 4 | 2
Extremity Necrosis (Vascular disorders) | 3 | 0
Femoral Artery Occlusion (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 4 | 1
Hypertensive Crisis (Vascular disorders) | 3 | 2
Hypertensive Emergency (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 2 | 2
Intermittent Claudication (Vascular disorders) | 0 | 3
Orthostatic Hypotension (Vascular disorders) | 3 | 2
Peripheral Arterial Occlusive Disease (Vascular disorders) | 58 | 16
Peripheral Artery Dissection (Vascular disorders) | 9 | 2
Peripheral Artery Stenosis (Vascular disorders) | 58 | 35
Peripheral Artery Thrombosis (Vascular disorders) | 3 | 3
Peripheral Ischaemia (Vascular disorders) | 5 | 2
Varicose Vein (Vascular disorders) | 0 | 1
Vascular Insufficiency (Vascular disorders) | 1 | 0
Vasospasm (Vascular disorders) | 3 | 2
Venous Insufficiency (Vascular disorders) | 0 | 2
Venous Thrombosis (Vascular disorders) | 1 | 0
Vessel Perforation (Vascular disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Acute Ischemia Left Lower Leg (General disorders) | 0 | 1 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Admission to Psychiatry (General disorders) | 1 | 0 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Chest Pain Syndrome with Acute Moderate Pericardia (General disorders) | 1 | 0 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Claudication Left Leg (General disorders) | 0 | 1 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Gangrene on Left Great Toe (General disorders) | 0 | 1 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
I & D with Partial Left Hallux Amputation (General disorders) | 0 | 1 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Occluded Left Sfa Stent (General disorders) | 1 | 0 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Occlusion of Right At & Dp (General disorders) | 1 | 0 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Occlusion of Left At and Stenosis of Left Tpt (General disorders) | 0 | 1 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Profundus Stenosis (General disorders) | 1 | 0 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
Ulcerated Basalioma Left Eyelid (General disorders) | 1 | 0 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lutonix DCB (N=287) | Standard Balloon Angioplasty Catheter (N=155)
Gangrene (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 3 | 3
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 4 | 5
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Embolism Arterial (Vascular disorders) | 6 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 6 | 1
Peripheral Artery Dissection (Vascular disorders) | 6 | 1
Peripheral Artery Stenosis (Vascular disorders) | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 1
Vasospasm (Vascular disorders) | 8 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 | 0
Local Swelling (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 2 | 1
Puncture Site Haemorrhage (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 1
Stent Malfunction (General disorders) | 0 | 1
Vessel Puncture Site Haematoma (General disorders) | 7 | 2
Arthritis Bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 1 | 1
Localised Infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 2 | 1
Incision Site Complication (Injury, poisoning and procedural complications) | 2 | 0
Peripheral Arterial Reocclusion (Injury, poisoning and procedural complications) | 3 | 2
Peripheral Artery Restenosis (Injury, poisoning and procedural complications) | 3 | 4
Scrotal Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 5 | 3
Wound (Injury, poisoning and procedural complications) | 0 | 3
Haemoglobin Decreased (Investigations) | 1 | 0
Urine Analysis Abnormal (Investigations) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephropathy Toxic (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriovenous Fistula (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 4 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 7 | 1
Peripheral Artery Dissection (Vascular disorders) | 10 | 2
Vasospasm (Vascular disorders) | 11 | 4
Vessel Perforation (Vascular disorders) | 1 | 0
Worsening of Peripheral Artery Disease (General disorders) | 0 | 2 — This SAE was uncoded in terms of Organ System in the Clinical Study Report and therefore, is added here under "General Disorders".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT01870401/Prot_SAP_000.pdf